CLINICAL TRIAL: NCT04168437
Title: Optimizing Chronic Pain Management Through Patient Engagement With Quality of Life Measures: A Randomized Controlled Trial
Brief Title: Optimizing Chronic Pain Management Through Patient Engagement With Quality of Life Measures
Acronym: OPTIQUAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Texas Health Science Center (Other)
Responsible Party: Principal Investigator, John C. Licciardone, D.O., M.S., M.B.A., Principal Investigator, University of North Texas Health Science Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-169
Record Dates: First submitted 2019-11-15; First posted 2019-11-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Chronic Low Back Pain
Keywords: Back Pain; Quality of Life; PROMIS-29; PRECISION Pain Research Registry
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health-Related Quality of Life Report (Experimental): Participants randomized to this arm will receive the 2- page Health-Related Quality of Life Report.
  Interventions: Other: Health-Related Quality of Life Report
- Wait List to Receive the Report (No Intervention): Participants randomized to this arm will receive the 2- page Health-Related Quality of Life Report following completion of the study.

INTERVENTIONS:
Other: Health-Related Quality of Life Report — Two page report and interpretation guide based on SPADE cluster scores
  Arms: Health-Related Quality of Life Report

SUMMARY:
This study evaluates the use of a health-related quality of life report based on the SPADE cluster (sleep disturbance, pain interference with activities, anxiety, depression, and low energy/fatigue) derived from the PROMIS-29 instrument in patients with chronic low back pain. Half of the participants will receive the report, while the other half will not.

DETAILED DESCRIPTION:
The health-related quality of life report provides participants with an overall score on the SPADE cluster and scores on each of its five component scales. The recently released Federal Pain Research Strategy states that pain cannot be measured in isolation, but rather should be assessed in conjunction with other outcome measures in 'non-pain domains,' such as quality of life. It recognizes that pain may be affected by, and affect, such patient attributes as sleep, mood, cognition, function, and quality of life. Further, the report states that improvement in pain without concomitant improvement in other domains may not constitute a clinically meaningful outcome. This study primarily aims to assess the utility of a health-related quality of life report in improving quality of life, back pain intensity, and back-related disability in participants with chronic low back pain. Another aspect of the study will be to determine how the health-related quality of life report may impact the physician-patient interaction. This will be assessed using validated measures of physician interpersonal manner, empathy, and communication style, as well as end-of-trial survey data acquired from participants assigned to the experimental group. The survey will include an overall assessment of the report, as well as specific actions attributed to the report.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Low Back Pain AND SPADE Cluster Score ≥ 55

Exclusion Criteria:

* Absence of Chronic Low Back Pain OR SPADE Cluster Score < 55

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
PROMIS-29 Quality of Life Measures | 3 Months Post-Randomization
  SPADE Cluster Scores (population mean, 50)

SECONDARY OUTCOMES:
Low Back Pain Intensity | 3 Months Post-Randomization
  Numerical Rating Scale for Pain (0-10)
Back-Related Disability | 3 Months Post-Randomization
  Roland-Morris Disability Questionnaire (0-24)

CONTACTS AND LOCATIONS:
Overall Officials: John C Licciardone, DO, MS, MBA, Principal Investigator — University of North Texas Health Science Center
Locations (1):
- University of North Texas Health Science Center, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No